CLINICAL TRIAL: NCT02945670
Title: Using Focus Group to Explore Cultural Acceptability of Long Acting Contraception in a Diverse, Urban Population.
Brief Title: Using Focus Group to Explore Cultural Acceptability of Contraception
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jeannette E. South-Paul, Andrew W. Mathieson UPMC Professor and Chair, University of Pittsburgh
Other Study IDs: Merck IIS# 55000
Record Dates: First submitted 2016-10-23; First posted 2016-10-26 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Contraception
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Focus Group — We had recruited 64 women and completed 7 focus group sessions

SUMMARY:
The purpose of this study is to learn what women of childbearing age think of Long Acting Reversible Contraception. A variety of myths regarding LARCs have been described in the literature. This study is designed to asses women's cultural belief's regarding LARCs. Investigators are looking to collect information from women in general, rather than solely who are seeking contraception. Investigators will be recruiting women ages 18-45 years from seven family health centers affiliated with UPMC. Participants will be asked to a attend a 60-90 minutes focus group session. During the session the facilitator will try to engage participants in a discussion about contraception in general. They will also be asked to complete a short demographic survey of 8-12 questions. Data from focus groups will be assessed for recurring themes which will be used to create a cultural survey instrument that will be used in the second phase of the study.

DETAILED DESCRIPTION:
Following approval by the University of Pittsburgh institutional review board (IRB), female participants between 18 and 45 years of age seeking care for contraception or other women's health services were recruited from seven Family Health Centers (FHCs) partnered with the Department of Family Medicine. The participants agreed to participate in one 2 hour facilitated focus group session (recorded for later transcription) to discuss their perceptions about contraception.

Recordings were transcribed and de-identified. The resulting texts were coded by a team. Concepts and themes that arose from the coding were analyzed to inform the development of a survey on the topic of perspectives on contraception.

Qualitative analysis of the transcripts and coding was carried out and results were shared in pubic fora.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-45 years
* Not pregnant

Exclusion Criteria:

* Pregnancy
* Male

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women age 18-45 years and not pregnant at the time of enrollment
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Level of acceptance of contraception among diverse women | Three months
  Level of acceptance: 1-Totally not accepted 2-May accept 3-Neither accept/not accept 4-Accept with preservation 5-Totally accept

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette E. South-Paul, MD, Principal Investigator — University of Pittsburgh
Locations (7):
- United States (7):
  - Latterman Family Health Center, McKeesport, Pennsylvania
  - New Kensington Family Health Center, New Kensington, Pennsylvania
  - UPMC Matilda Theiss Health Center, Pittsburgh, Pennsylvania
  - Squirrel Hill Family Practice, Pittsburgh, Pennsylvania
  - UPMC Bloomfiled-Garfield FHC, Pittsburgh, Pennsylvania
  - Lawrenceville Family Health Center, Pittsburgh, Pennsylvania
  - Shadyside Family Health Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mestad R, Secura G, Allsworth JE, Madden T, Zhao Q, Peipert JF. Acceptance of long-acting reversible contraceptive methods by adolescent participants in the Contraceptive CHOICE Project. Contraception. 2011 Nov;84(5):493-8. doi: 10.1016/j.contraception.2011.03.001. Epub 2011 Apr 27. PMID 22018123
- [Background] Secura GM, Allsworth JE, Madden T, Mullersman JL, Peipert JF. The Contraceptive CHOICE Project: reducing barriers to long-acting reversible contraception. Am J Obstet Gynecol. 2010 Aug;203(2):115.e1-7. doi: 10.1016/j.ajog.2010.04.017. Epub 2010 Jun 11. PMID 20541171
- [Background] Romero L, Pazol K, Warner L, Gavin L, Moskosky S, Besera G, Loyola Briceno AC, Jatlaoui T, Barfield W; Centers for Disease Control and Prevention (CDC). Vital signs: trends in use of long-acting reversible contraception among teens aged 15-19 years seeking contraceptive services-United States, 2005-2013. MMWR Morb Mortal Wkly Rep. 2015 Apr 10;64(13):363-9. PMID 25856258
- [Background] Harper CC, Blum M, de Bocanegra HT, Darney PD, Speidel JJ, Policar M, Drey EA. Challenges in translating evidence to practice: the provision of intrauterine contraception. Obstet Gynecol. 2008 Jun;111(6):1359-69. doi: 10.1097/AOG.0b013e318173fd83. PMID 18515520
- [Background] Stanwood NL, Bradley KA. Young pregnant women's knowledge of modern intrauterine devices. Obstet Gynecol. 2006 Dec;108(6):1417-22. doi: 10.1097/01.AOG.0000245447.56585.a0. PMID 17138775
- [Background] Whitaker AK, Sisco KM, Tomlinson AN, Dude AM, Martins SL. Use of the intrauterine device among adolescent and young adult women in the United States from 2002 to 2010. J Adolesc Health. 2013 Sep;53(3):401-6. doi: 10.1016/j.jadohealth.2013.04.011. Epub 2013 Jun 12. PMID 23763968
- [Background] Damle LF, Gohari AC, McEvoy AK, Desale SY, Gomez-Lobo V. Early initiation of postpartum contraception: does it decrease rapid repeat pregnancy in adolescents? J Pediatr Adolesc Gynecol. 2015 Feb;28(1):57-62. doi: 10.1016/j.jpag.2014.04.005. Epub 2014 May 5. PMID 25555302
- [Background] Okpo E, Allerton L, Brechin S. 'But you can't reverse a hysterectomy!' Perceptions of long acting reversible contraception (LARC) among young women aged 16-24 years: a qualitative study. Public Health. 2014 Oct;128(10):934-9. doi: 10.1016/j.puhe.2014.08.012. Epub 2014 Oct 22. PMID 25369357
- [Background] Greenberg KB, Makino KK, Coles MS. Factors associated with provision of long-acting reversible contraception among adolescent health care providers. J Adolesc Health. 2013 Mar;52(3):372-4. doi: 10.1016/j.jadohealth.2012.11.003. PMID 23427785
- [Background] Rubin SE, Davis K, McKee MD. New york city physicians' views of providing long-acting reversible contraception to adolescents. Ann Fam Med. 2013 Mar-Apr;11(2):130-6. doi: 10.1370/afm.1450. PMID 23508599
- [Background] Russo JA, Miller E, Gold MA. Myths and misconceptions about long-acting reversible contraception (LARC). J Adolesc Health. 2013 Apr;52(4 Suppl):S14-21. doi: 10.1016/j.jadohealth.2013.02.003. PMID 23535052
- [Background] Roncancio AM, Ward KK, Berenson AB. The use of effective contraception among young Hispanic women: the role of acculturation. J Pediatr Adolesc Gynecol. 2012 Feb;25(1):35-8. doi: 10.1016/j.jpag.2011.08.008. Epub 2011 Nov 3. PMID 22051784
- [Background] Doescher MP, Saver BG, Franks P, Fiscella K. Racial and ethnic disparities in perceptions of physician style and trust. Arch Fam Med. 2000 Nov-Dec;9(10):1156-63. doi: 10.1001/archfami.9.10.1156. PMID 11115223
- [Background] Kissling E, Valenciano M, Larrauri A, Oroszi B, Cohen JM, Nunes B, Pitigoi D, Rizzo C, Rebolledo J, Paradowska-Stankiewicz I, Jimenez-Jorge S, Horvath JK, Daviaud I, Guiomar R, Necula G, Bella A, O'Donnell J, Gluchowska M, Ciancio BC, Nicoll A, Moren A. Low and decreasing vaccine effectiveness against influenza A(H3) in 2011/12 among vaccination target groups in Europe: results from the I-MOVE multicentre case-control study. Euro Surveill. 2013 Jan 31;18(5):20390. doi: 10.2807/ese.18.05.20390-en. PMID 23399425
- [Result] Lin C, South-Paul JE, Maier JS, deBorja L, Al Aaraj Y, Burley C, Mena J,.Using Focus Group to Explore Cultural Acceptability of Long Acting Contraception in a Diverse, Urban Population. North American Primary Care Research Group Annual Meeting - NOV 2017 / Montreal, QB (https://www.napcrg.org/conferences/43/sessions/20937)
- [Result] Cuddeback M, Ifthikhar R, Narayanan A. Assessment of Cultural Acceptability of Long Acting Reversible Contraception in a Diverse, Urban Population. North American Primary Care Research Group Annual Meeting - Toronto, ON / NOV. 2019. (https://www.napcrg.org/conferences/2001/sessions/770)